CLINICAL TRIAL: NCT01762657
Title: A Phase 3, Randomized, Double-Blind, Multinational, Placebo-Controlled Study to Evaluate the Safety and Efficacy in Diminishing Insulin Requirements Utilizing Oral Cyclosporine With Oral Lansoprazole in Children and Adults With Existing Type 1 Diabetes Mellitus
Brief Title: The Insulin Independence Trial (IIT) Evaluating the Safety and Efficacy of Oral Cyclosporine and Oral Lansoprazole for Insulin Independence Among Patients With Existing Type 1 Diabetes
Acronym: IIT
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study stopped prior to Patient Enrollment
Sponsor: Perle Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Perle-1102
Record Dates: First submitted 2013-01-02; First posted 2013-01-08 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Insulin Independence; Beta Regeneration; Immune Tolerance Agent; Lanzoprazole; Cyclosporine
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Cyclosporine; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral CyclosporineA and Oral Lansoprazole (Experimental): Oral Cyclosporine A dosed at 7.5 mg/kg/day in two divided dosages given with Lansoprazole dosed at 30 mg per day in two divided dosages for subjects aged 8-15 year and 60 mg per day for those aged 16-60.
  Interventions: Drug: Oral Cyclosporine and Oral Lansoprazole
- Placebos (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Oral Cyclosporine and Oral Lansoprazole — Oral Cyclosporine A dosed at 7.5 mg/kg/day and Oral Lansoprazole dosed at 30 mg in two divided dosages to subjects ages 8-15 and 60 60 mg in divided dosages to subjects ages 16-60. The Cyclosporine A and Lansoprazole may be given as an oral tablet/capsule or oral suspension.
  Arms: Oral CyclosporineA and Oral Lansoprazole
Drug: Placebos — Two oral placebos are given at breakfast and dinner. The placebos may be given as an oral tablets/capsules or oral suspensions.
  Arms: Placebos

SUMMARY:
The purpose of this study is to determine if oral Cyclosporine A and oral Lansoprazole are effective in rendering patients with existing type 1 diabetes, insulin independent. This two-arm study was designed to evaluate the safety and efficacy for insulin independence by utilizing the FDA-approved oral immune tolerance agent, Cyclosporine A, and the FDA-approved proton-pump inhibitor, Lansoprazole. Lansoprazole and other proton-pump inhibitors increase gastrin levels. Gastrin was initially shown to have the potential to increase new beta cell formation in 1955 (Zollinger RM and Ellison EH. Ann Surg. 1955;142(4):709-23).

Studies with the immune tolerance agent, Cyclosporine A, previously demonstrated that among recently diagnosed type 1 diabetes patients, insulin independence was achieved in as many as 67.5% of patients within 7 weeks of therapy (Bougneres PF et al. N Engl J Med. 1988:17;318(11):663-70). Cyclosporine A protected the remaining beta cells from further autoimmune attack, but over time, there was limited beta cell regeneration, and insulin was ultimately required by all patients. Therefore, this study proposes the usage of Cyclosporine A with a beta regeneration agent.

Follow-up studies for up to 13 years among 285 type 1 patients utilizing Cyclosporine A for 20 months, did not demonstrate renal or other side effects (Assan R. et al. Diabetes Metab Res Rev. 2002;18(6):464-72). Human clinical trials with gastrin and epidermal growth factor demonstrated reductions in daily insulin requirements by much as 75% within 3 months following four weeks of therapy among existing type 1 diabetes patients (Transition Therapeutics, March 5, 2007 http://www.transitiontherapeutics.com/media/archive.php Accessed January 1, 2013). Lack of the ability to sustain these results was likely due to the ongoing autoimmune attack on the new beta cells generated by therapy. Gastrin alone has been shown to induce beta cell neogenesis from human pancreatic ductal tissue without epidermal growth factor in in vitro studies (Suarez-Pinzon WL et al. JCEM. 2005;90(6):3401-3409).

Type 1 diabetes is an autoimmune disease. Despite evidence that many different immune tolerance agents have successfully reversed diabetes in rodent type 1 models, none have been successful in sustaining insulin independence in man (Ablamunits V et al. Ann NY Acad Sci. 2007;1103:19-32). The distinctions and complexities of islets in man are far different than that of rodents (Levetan CS and Pierce SM. Endocr Pract. 2012 Nov 27:1-36 Epub ahead of print). We hypothesize that in man, both an immune tolerance agent and a beta regeneration agent are required to sustain insulin independence.

Based upon proton-pump inhibitors having been shown to increase plasma gastrin levels up to 10-fold, this clinical trial utilizes the oral proton-pump inhibitor, Lansoprazole. This study will determine the safety and efficacy of Cyclosporine A used with and without Lansoprazole to determine the impact on insulin independence among patients with existing type 1 diabetes.

Cyclosporine A is utilized to protect the new beta cells formed by Lansoprazole. The combination of the two therapies may render reductions in insulin requirements and have a greater impact on sustained insulin independence than previously reported with Cyclosporine A or gastrin alone among type 1 patients.A

This 52-week study consists of two treatment arms designed to assess the safety and efficacy of achieving insulin independence using:

* Oral Lansoprazole/Oral Cyclosporine A
* Oral Placebo/Oral Placebo

It is hypothesized that the combination of oral Cyclosporine A and oral Lansoprazole will safely render significantly more patients with existing type 1 diabetes, insulin independent and may serve as a novel and innovative treatment approach for patients with type 1 diabetes utilizing two FDA-approved therapies.

ELIGIBILITY:
Inclusion Criteria:

1. They are male or female, 8-60 years of age
2. They have a history of onset of type 1 Diabetes Mellitus at or before 20 years of age; or have documentation of autoimmunity testing to the pancreas to include one of more of the following tests

   * Islet-cell autoantibodies 512 (ICA512)/islet antigen-2 (IA-2),
   * Glutamic Acid Decarboxylase (GAD) autoantibodies, or
   * Insulin autoantibodies (in subjects on insulin for more than 2 weeks, ICA512/IA-2 or GAD must be positive)
3. They have a C-peptide of greater than or equal to to 0.6 ng/mL (0.2 nmol/L)
4. They have a Hemoglobin A1C levels of less than 9%
5. They are able and willing to participate in the study, as evidenced by providing written informed consent
6. Females must be post-menopausal (at least 1 year without spontaneous menses) or surgically sterile (tubal ligation or hysterectomy at least 6 months prior to enrollment), or to have a negative pregnancy test and practice acceptable contraception [e.g., oral, intramuscular, or implanted hormonal contraception, sexual partner with nonreversed vasectomy (with azoospermia in 2 tests), 2 barrier methods (e.g., condom, diaphragm, or spermicide), or intrauterine device]. Females of childbearing potential must undergo pregnancy testing within 24 hours prior to administration of the first dose of study drug.

Exclusion Criteria:

1. Prior administration of immune tolerance therapy or immune tolerance clinical trial for type 1 diabetes
2. Participation in any type of therapeutic drug or vaccine clinical trial within the last 12 weeks before randomization at Study Day 0
3. Any medical condition that, in the opinion of the investigator, would interfere with safe completion of the trial
4. Pregnant females or lactating females who intend to provide their own breast milk to the baby during the study
5. Current therapy with GLP-1 receptor agonists (e.g., exenatide or pramlintide), or any other agents that might stimulate pancreatic beta cell regeneration or insulin secretion
6. Current treatment with oral antidiabetic agents
7. Evidence of active or latent tuberculosis
8. Vaccination with a live virus or organism within the 8 weeks before randomization continuing through week 52 of the study

   * Influenza vaccination with a killed virus, including booster vaccinations, within 4 weeks before or after each dosing cycle
   * Vaccination with other antigens or killed organisms within 8 weeks before or after each dosing cycle
9. Systolic or diastolic blood pressure >150 mmHg and 90 mmHg, respectively, as measured by an appropriately sized cuff;
10. A body mass index (BMI) >28 kg/m2
11. Worsening retinopathy, angina, or congestive heart failure
12. A history or presence of acute or chronic pancreatitis
13. A history or presence of any illness, disease, or condition that could impact patient safety or evaluability of drug effect, in the Investigator's opinion
14. An episode of severe hypoglycemia (defined as a change in mental status requiring assistance) during the prior 30 days
15. An episode of diabetic ketoacidosis during the prior 6 months
16. Received any new hypoglycemic medications within the past 3 months
17. An aspartate transaminase (AST), alanine transaminase (ALT), or total bilirubin level >2 times the upper limit of normal (ULN)
18. A blood urea nitrogen (BUN) level >50 mg/dL or a serum creatinine level >1.4 mg/dL
19. A serum amylase level >1.5 times the ULN or a serum lipase level >2 times the ULN
20. A history of substance abuse or dependence in the past year as defined by the Diagnostic and Statistical Manual of Mental Disorders, (DSM V) criteria

Ages: 8 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Insulin Requirements Among Patients Treated with Oral Cyclosporine and Oral Lansoprazole | 26 and 52 weeks

SECONDARY OUTCOMES:
Glucagon C-peptide (under the curve) and Hemoglobin A1C levels among patients with existing type 1 diabetes treated with Cyclosporine and Lansoprazole | 26 and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Claresa Levetan, MD, Principal Investigator — Perle Bioscience, Inc.

REFERENCES:
- [Background] Assan R, Blanchet F, Feutren G, Timsit J, Larger E, Boitard C, Amiel C, Bach JF. Normal renal function 8 to 13 years after cyclosporin A therapy in 285 diabetic patients. Diabetes Metab Res Rev. 2002 Nov-Dec;18(6):464-72. doi: 10.1002/dmrr.325. PMID 12469360
- [Background] Bougneres PF, Carel JC, Castano L, Boitard C, Gardin JP, Landais P, Hors J, Mihatsch MJ, Paillard M, Chaussain JL, et al. Factors associated with early remission of type I diabetes in children treated with cyclosporine. N Engl J Med. 1988 Mar 17;318(11):663-70. doi: 10.1056/NEJM198803173181103. PMID 3125434
- [Background] Wang TC, Bonner-Weir S, Oates PS, Chulak M, Simon B, Merlino GT, Schmidt EV, Brand SJ. Pancreatic gastrin stimulates islet differentiation of transforming growth factor alpha-induced ductular precursor cells. J Clin Invest. 1993 Sep;92(3):1349-56. doi: 10.1172/JCI116708. PMID 8376589
- See also: MedlinePlus related topics: Diabetes Diabetes Medicines Diabetes Type 1 — http://www.nlm.nih.gov/medlineplus/diabetestype1.html